CLINICAL TRIAL: NCT02268006
Title: Preoperative Radiochemotherapy With IMRT - Simultaneous Integrated Boost in Locally Advanced Rectal Cancer - BISER
Brief Title: IMRT-SIB and Capecitabine in Preoperative Rectal Cancer Treatment
Acronym: BISER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 41/12/13
Record Dates: First submitted 2014-02-02; First posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-09

CONDITIONS: Rectal Carcinoma
Keywords: rectal carcinoma; preoperative radiochemotherapy; IMRT; SIB
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Surgical Procedures, Operative

ARMS (1):
- IMRT-SIB (Other)
  Interventions: Radiation: IMRT-SIB; Drug: Capecitabine; Procedure: Surgery

INTERVENTIONS:
Radiation: IMRT-SIB
Drug: Capecitabine
  Other Names: (Xeloda, Capecitabine Teva, Ecansya)
Procedure: Surgery
  Other Names: Total Mesorectal Exscision

SUMMARY:
RATIONALE: Using small radiation beamlets of different intensity, IMRT (intensity modulated radiation therapy) allows shaping the dose around planning target volume with better sparing of normal tissue comparing to 3D conformal radiotherapy. It allows daily delivery of higher dose to the tumor with simultaneous integrated boost (SIB), consequently shortening total treatment time with potentially better response to treatment. In advanced rectal adenocarcinoma excellent response to preoperative radiochemotherapy with complete eradication of the primary tumor observed in the histopathological specimen (pathological complete response, pCR) correlates with a favorable overall prognosis, so trying to achieve better response to preoperative treatment with higher pCR seams feasible.

PURPOSE:The hypothesis of this study is that in preoperative radiochemotherapy for locally advanced rectal adenocarcinoma shortening of the total treatment time with IMRT-SIB to 22 daily fractions concomitant with capecitabine results in an improved pCR rate from 9% (Slovenian trial) to 25%. Secondary objectives are to evaluate pathological down-staging rate, histopathological R0 resection rate, sphincter preservation rate, perioperative surgical complication rate, local control, disease-free survival (DFS), overall survival (OS), late toxicity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven newly diagnosed primary rectal adenocarcinoma
* Locally advanced tumor fulfilling at least one of the following criteria on pelvic MRI:

  * T ≥ 3 or
  * N ≥ 1
  * Positive mesorectal fascia (MRF), i.e. tumor or lymph node one mm or less from the mesorectal fascia
  * Tumor located od 0 - 15 cm above anocutaneous junction or below peritoneum
* Age 18 years and more
* Signed informed consent
* WHO Performance Status 0-2
* Patients is considered to be mentally and physically ft for chemotherapy as judged by oncologist
* Adequate hematological, hepatic and renal function (WBC ≥ 3.0 x 109/L, neu ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, renal clearance ≥ 50 ml/min, bilirubin ≤ 3x normal value, aspartate transaminase/alanine transaminase (AST/ALT) ≤ 2,5x normal value)

Exclusion Criteria:

* T4 inoperable tumor - extensive growth into cranial part of the sacrum (above S3) or the lumbosacral nerve roots
* Metastatic or recurrent rectal cancer
* Other co-existing malignancy or malignancy within the past 5 years, with the exception of adequately treated in situ carcinoma of the cervix or basal cell carcinoma of the skin
* Chronic bowel inflammatory disease
* Pregnant or lactating patient
* Significant heart disease (uncontrolled hypertension despite of medication (> 150/100 mmHg), New York Heart Association (NYHA) class III or IV heart disease,unstable angina or myocardial infarction within the past 1 year prior the study entry, history of significant ventricular arrhythmia requiring treatment)
* Inability to consciously sign the consent form due to physical or psychological disabilities

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission rate (pCR) | after the pathological examination of surgical specimens i.e. within 14 days after the operation

SECONDARY OUTCOMES:
Toxicity | According to NCI-CTC (version 4.0): every week for 16 week preoperative, perioperative (0-30 days postoperative), early (30 days - 6 months postoperative), and late (more than 6 months postoperative)
Histopathological R0 resection rate | after the pathological examination of resected specimens i.e. within 14 days after the operation
Tumor down-staging rate | after the pathological examination of resected specimens i.e. within 14 days after the operation
Rate of sphincter sparing surgical procedure | Toxicity/safety: one month after surgery.
Loco-regional failure rate | after 3y and 5y of operation
Disease-free survival | after 3y and 5y of operation
Overall survival | after 3y and 5y of the operation
Quality of life | before the treatment, after surgery, after1,2,3,4 and 5 years of the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology, Ljubljana, Slovenia

REFERENCES:
- [Background] Engels B, De Ridder M, Tournel K, Sermeus A, De Coninck P, Verellen D, Storme GA. Preoperative helical tomotherapy and megavoltage computed tomography for rectal cancer: impact on the irradiated volume of small bowel. Int J Radiat Oncol Biol Phys. 2009 Aug 1;74(5):1476-80. doi: 10.1016/j.ijrobp.2008.10.017. Epub 2009 Feb 21. PMID 19231097
- [Background] Arbea L, Ramos LI, Martinez-Monge R, Moreno M, Aristu J. Intensity-modulated radiation therapy (IMRT) vs. 3D conformal radiotherapy (3DCRT) in locally advanced rectal cancer (LARC): dosimetric comparison and clinical implications. Radiat Oncol. 2010 Feb 26;5:17. doi: 10.1186/1748-717X-5-17. PMID 20187944
- [Background] Mok H, Crane CH, Palmer MB, Briere TM, Beddar S, Delclos ME, Krishnan S, Das P. Intensity modulated radiation therapy (IMRT): differences in target volumes and improvement in clinically relevant doses to small bowel in rectal carcinoma. Radiat Oncol. 2011 Jun 8;6:63. doi: 10.1186/1748-717X-6-63. PMID 21651775
- [Background] Li JL, Ji JF, Cai Y, Li XF, Li YH, Wu H, Xu B, Dou FY, Li ZY, Bu ZD, Wu AW, Tham IW. Preoperative concomitant boost intensity-modulated radiotherapy with oral capecitabine in locally advanced mid-low rectal cancer: a phase II trial. Radiother Oncol. 2012 Jan;102(1):4-9. doi: 10.1016/j.radonc.2011.07.030. Epub 2011 Sep 6. PMID 21903285
- [Result] Velenik V, Anderluh F, Oblak I, Strojan P, Zakotnik B. Capecitabine as a radiosensitizing agent in neoadjuvant treatment of locally advanced resectable rectal cancer: prospective phase II trial. Croat Med J. 2006 Oct;47(5):693-700. PMID 17042060
- [Result] Velenik V, Oblak I, Anderluh F. Long-term results from a randomized phase II trial of neoadjuvant combined-modality therapy for locally advanced rectal cancer. Radiat Oncol. 2010 Sep 29;5:88. doi: 10.1186/1748-717X-5-88. PMID 20920276